CLINICAL TRIAL: NCT03072628
Title: The Effects of Electronic Cigarettes on Endothelial Function and Oxidative Stress
Brief Title: E-cigarettes, Nicotine Inhaler, and Blood Vessel Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Holly R Middlekauff, Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 14-000743-AM-00008
Record Dates: First submitted 2017-03-02; First posted 2017-03-07 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Nicotine Dependence
Keywords: nicotine; sympathetic nerve activity; oxidative stress
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Electronic Nicotine Delivery Systems; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Nicotine: use e-cig with nicotine (Experimental): One time exposure to e-cig with nicotine
  Interventions: Other: e-cig with nicotine
- no nicotine: use e-cig without nicotine (Experimental): One time exposure to e-cig without nicotine
  Interventions: Other: e-cig without nicotine
- Nicotine inhaler: use a nictoine inhaler (Experimental): One time exposure to nicotine inhaler
  Interventions: Other: nicotine inhaler
- Sham control (Sham Comparator): Use an empty e-cigarette
  Interventions: Other: sham control

INTERVENTIONS:
Other: e-cig with nicotine — use an e-cig with nicotine for 30 minutes
  Arms: Nicotine: use e-cig with nicotine
Other: e-cig without nicotine — use an e-cig without nicotine for 30 minutes
  Arms: no nicotine: use e-cig without nicotine
Other: nicotine inhaler — use a nicotine inhaler for 30 minutes
  Arms: Nicotine inhaler: use a nictoine inhaler
Other: sham control — use an empty e-cigarette for 30 minutes
  Arms: Sham control

SUMMARY:
Randomized controlled trial of electronic cigarettes with nicotine, without nicotine, nicotine inhaler, and sham-control on endothelial function, oxidative stress and sympathetic nerve activity

DETAILED DESCRIPTION:
Participants will have an acute exposure on 4 occasions1) e-cigarette with nicotine, 2) e-cigarette without nicotine, 3) nicotine inhaler, 4) sham control and undergo ECG recording for heart rate variability, endothelial function measurement using ultrasound ("FMD") and blood tests for oxidative stress markers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy

Exclusion Criteria:

* Cardiac disease
* Respiratory disease
* Diabetes mellitus

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 148 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Flow Mediated dilatation (FMD) | 10 minutes after exposure
  FMD is a measure of endothelial function
Heart rate variability (HRV) | 10 minutes after exposure
  HRV is a measure of cardiac sympathetic tone

SECONDARY OUTCOMES:
Paraoxonase (PON) | ~30 minutes after exposure
  PON is a measure of oxidative stress

CONTACTS AND LOCATIONS:
Locations (1):
- UCaliforniaLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No